CLINICAL TRIAL: NCT03237429
Title: The Relationship Between Volemic Status as Assessed by Bioimpedance Spectroscopy, Arterial Stiffness and Hemodynamic Instability During Induction of General Anesthesia
Brief Title: The Relationship Between BCM, Arterial Stiffness and Hemodynamic Instability During Induction of General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, Professor, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: GTPopaUMP
Record Dates: First submitted 2017-07-30; First posted 2017-08-02 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Vascular Stiffness; Hypotension on Induction; Anesthesia; Reaction
Keywords: bioimpedance spectroscopy; arterial stiffness
MeSH Terms: interventions — Carotid-Femoral Pulse Wave Velocity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cancer patients: The first study population will represent patients scheduled for surgery for a new diagnosed cancer pathology
  Interventions: Diagnostic Test: bioimpedance spectroscopy
- non-cancer patients: The second study population will represent patients scheduled for surgery not for cancer disease
  Interventions: Diagnostic Test: bioimpedance spectroscopy

INTERVENTIONS:
Diagnostic Test: bioimpedance spectroscopy — Bioimpedance spectroscopy-The technique involves attaching electrodes to the patient's forearm and ipsilateral ankle, with the patient in a supine position. The BCM measures the body resistance and reactance to electrical currents of 50 discrete frequencies, ranging between 5 and 1000 kHz. Based on a fluid model using these resistances, the extracellular water (ECW), the intracellular water (ICW) and the total body water (TBW) are calculated. These volumes are then used to determine the amount of fluid.
  Carotid-femoral pulse wave velocity-will be determined by arterial applanation tonometry using the Sphygmocor system by sequentially recording ECG-gated carotid and femoral artery waveforms.. Pulse wave signals will be recorded by tonometers positioned at the base of the right common carotid artery and over the right femoral artery.
  Other Names: Carotid-femoral pulse wave velocity

SUMMARY:
Arterial hypotension during induction of general anesthesia is a risk factor for developing postoperative cardiovascular complications. After induction of general anesthesia patients have a high risk of developing arterial hypotension due to anesthetic drugs who can depress cardiac contractility and determine vasodilatation. Previous studies have shown that even short periods of hypotension with a mean arterial pressure of less than 55 mmHg during surgery is associated with an increased incidence of cardiac injury and acute kidney injury in the postoperative period.

The volemic status of the patients in the preoperative period is very difficult to quantify and can vary due to comorbidities of the patient, chronic treatment, preoperative fasting. Bioimpedance is recognized by over 30 years as a simple and non invasive technique to determine the volemic status especially in the hemodialysed patients. A new device BCM- Body Composition Monitoring (Fresenius Medical Care) offers a simple method to determine extracellular water and total body water. These volumes are determined by measuring impedance at 50 different frequencies thru electrodes placed at the ankle and wrist. BCM can also determine lean tissue mass and adipose tissue mass.

Increasing arterial stiffness is the main characteristic of arterial aging; this increase determines the increase of the afterload, left ventricular hypertrophy, the decrease of coronary and tissue perfusion. Arterial applanation tonometry is a non-invasive technique that has been shown to reliably provide indices of arterial stiffness.

In this study investigators wish to determine if there is a correlation between the hidric status determined by BCM, carotid-femural pulse wave velocity determined with SphygmoCor system and the development of hypotension during induction of general anesthesia. The measurements will be obtained before induction of general anesthesia in the pre-surgical area. During induction of general anesthesia with standard induction agents and Bispectral index monitoring, brachial blood pressure will be measured by a cuff every minute after the loss of verbal contact with the patient up to ten minutes after tracheal intubation. A hypotensive response to anesthesia will be defined as a drop in mean arterial pressure below 55mmHg or a drop in mean arterial pressure with more than 40% than the base line value of the patient before the surgery.

Measurement of the hidric status and aortic stiffness may represent a valid indicator of the risk of hypotension during anesthesia induction.

DETAILED DESCRIPTION:
Arterial hypotension during induction of general anesthesia is a risk factor for developing postoperative cardiovascular complications. After induction of general anesthesia patients have a high risk of developing arterial hypotension due to anesthetic drugs who can depress cardiac contractility and determine vasodilatation. Risk factors associated with increased incidence of arterial hypotension at induction of general anesthesia are age > 50 years, ASA risk class III or IV, using high doses of propofol or fetanyl at induction. Previous studies have shown that even short periods of hypotension with a mean arterial pressure of less than 55 mmHg during surgery is associated with an increased incidence of cardiac injury and acute kidney injury in the postoperative period. Even if it is known that arterial hypotension is associated with increased incidence of postoperative complications, the inferior limit and duration of hypotension is not well defined. The volemic status of the patients in the preoperative period is very difficult to quantify and can vary due to comorbidities of the patient, chronic treatment, preoperative fasting. Bioimpedance is recognized by over 30 years as a simple and non invasive technique to determine the volemic status especially in the hemodialyzed patients. A new device BCM- Body Composition Monitoring (Fresenius Medical Care) offers a simple method to determine extracellular water and total body water. These volumes are determined by measuring impedance at 50 different frequencies thrue electrodes placed at the ankle and wrist. BCM can also determine lean tissue mass and adipose tissue mass.

Increasing arterial stiffness is the main characteristic of arterial aging; this increase determines the increase of the afterload, left ventricular hypertrophy, the decrease of coronary and tissue perfusion. Increased arterial stiffness is associated with altered ability of maintaining a normal arterial pressure during stress conditions; it is known the risk of orthostatic hypotension in older patients wits increased arterial stiffness Arterial applanation tonometry is asimple, non-invasive technique that has been shown to reliably provide indices of arterial stiffness. Measuring carotid-femural pulse wave velocity thrue applanation tonometry is considered the "gold standard" for measuring arterial stiffness.In this study carotid-femoral pulse wave velocity will be determined by applanation tonometry using the Sphygmocor system by sequentially recording ECG-gated carotid and femoral artery waveforms. Pulse wave signals will be recorded by tonometers positioned at the base of the right common carotid artery and over the right femoral artery.

In this study investigators wish to determine if there is a correlation between the hidric status determined by BCM, carotid-femural pulse wave velocity determined with SphygmoCor system and the development of hypotension during induction of general anesthesia. The measurements will be obtained before induction of general anesthesia in the pre-surgical area. During induction of general anesthesia with standard induction agents(fentanyl propofol, rocuronium) and Bispectral index monitoring, brachial blood pressure will be measured by a cuff every minute after the loss of verbal contact with the patient up to ten minutes after tracheal intubation. A hypotensive response to anesthesia will be defined as a drop in mean arterial pressure below 55mmHg or a drop in mean arterial pressure with more than 40% than the base line value of the patient before the surgery.

Study population : patients who are going under surgery. Inclusion criteria: there will be two study populations. The first study population will represent patients scheduled for surgery for a new diagnosed cancer pathology. The second study population will represent patients scheduled for surgery not for cancer disease. Exclusion criteria: diabetes (on insulin therapy), renal insufficiency (creatinine>2.0mg/dl), history of arterial bypass), history of carotid endoarterectomy, atrial fibrillation/flutter, history of ischemic stroke, transient ischemic attack, myocardial infarction or coronary revascularization (any type) within 6 months, known left main or 3-vessel coronary disease positive myocardial perfusion study without subsequent revascularization, heart failure (>3 NYHA) class 3, known left ventricle ejection fraction <30%, pulmonary hypertension (PA systolic >50mmHg), right ventricle dysfunction, sepsis, pregnancy, limb amputation.

ELIGIBILITY:
Inclusion Criteria:

- patients scheduled for surgery for a new diagnosed cancer pathology

Exclusion Criteria:

* diabetes (on insulin therapy),
* renal insufficiency (creatinine>2.0mg/dl),
* history of arterial bypass, carotid endoarterectomy,
* history of atrial fibrillation/flutter, ischemic stroke, transient ischemic attack, myocardial infarction or coronary revascularization (any type) within 6 months,
* known left main or 3-vessel coronary disease positive myocardial perfusion study without subsequent revascularization,
* heart failure (>3 NYHA) class 3, known left ventricle ejection fraction <30%, pulmonary hypertension (PA systolic >50mmHg), right ventricle dysfunction,
* sepsis,
* pregnancy,
* limb amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients scheduled for surgery for a new diagnosed cancer pathology
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between the hydric status determined by BCM and the development of hypotension during induction of general anesthesia | 2 years
  Correlation between the hydric status determined by BCM and the development of hypotension during induction of general anesthesia
Correlation between arterial stiffness and hypotension during induction of general anesthesia | 2 years
  Correlation between the carotid-femural pulse wave velocity determined with SphygmoCor system and the development of hypotension during induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrie Siriopol, MD, PhD, Study Chair — GRT POPA
Locations (1):
- Regional Institute of Oncology, Iasi, Iași, Romania